CLINICAL TRIAL: NCT02275702
Title: Randomized Study of Preoperative Dexamethasone for Quality of Recovery in VATS Lung Resection Patients
Acronym: APV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: APV-100
Record Dates: First submitted 2014-09-23; First posted 2014-10-27 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: Dexamethasone; Quality of recovery questionnaire; QoR-40; Lung cancer; Video-assisted thoracoscopic
MeSH Terms: conditions — Lung Neoplasms | interventions — Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Placebo Comparator): saline solution IV, bolus
  Interventions: Drug: Saline solution
- Group 2 (Active Comparator): 0,1mg/kg systemic dose of dexamethasone, bolus
  Interventions: Drug: Dexamethasone IV

INTERVENTIONS:
Drug: Dexamethasone IV — It will be administered at the induction of the anesthesia
  Other Names: Decadron
  Arms: Group 2
Drug: Saline solution
  Arms: Group 1

SUMMARY:
The proposed study is a randomized, double-blind, placebo-controlled evaluation if a small dose of IV dexamethasone during induction anesthesia in association to pre and postoperative intercostal nerve block, improves quality of recovery of thoracoscopic lung resection patients.

DETAILED DESCRIPTION:
This is a study composed by 2 groups of 50 patients undergoing VATS for lung cancer. All subjets will receive intraoperative intercostal nerve block with a maximum dose of 2 mg/kg of bupivacaine with epinephrine 1:200.000 at the beginning and at the end of procedure.

The control group will receive a bolus dose of dexamethasone (0.1 mg/kg) and the placebo group saline solution. The study drug or placebo will be administered at the time of anesthetic induction (approximately 30 minutes before surgical incision). Patients will be evaluated daily with the quality of recovery questionary, visual analogue pain and portable spirometry. And, the patients will have pulmonary lung function assessed by portable spirometry.

ELIGIBILITY:
Inclusion Criteria:

* resectable stage I and II lung cancer patients submitted to VATS
* american society of anesthesiology Classification (ASA) I or II

Exclusion Criteria:

* chronic pain;
* chronic analgesic consumption;
* severe renal or liver disease;
* endocrine or mental diseases;
* poorly controlled diabetes;
* allergy to bupivacaine;
* previous thoracotomy;
* systemic use of corticosteroids;
* morbid obesity;
* poor French comprehension precluding completion of the QoR-40 questionnaire;
* patient refusal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be postoperative quality of recovery measured by postoperative quality of recovery score 40 (QoR-40) global score. | During the hospital stay and 1 year later

SECONDARY OUTCOMES:
Time of analgesia between the final intercostal nerve block and the first patient-controlled analgesia (PCA) request; | During the hospital stay and 1 year later

OTHER OUTCOMES:
Correlation between pain with visual analog scale and lung function through spirometry test with forced expiratory volume at one second (FEV1) and diffusion capacity (DLCO) | During the hospital stay and 1 year later
Total opioid dose consumption in each group | During the hospital stay and 1 year later
Side-effect of dexamethasone in the stress response to surgery | During the hospital stay and 1 year later

CONTACTS AND LOCATIONS:
Overall Officials: Paula A. Ugalde, Medicin, Principal Investigator — Institut Universitaire de Cardilogie et Pneumologie de Québec, IUCPQ
Locations (2):
- Canada (2):
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, IUCPQ, Québec
  - IUCPQ, Québec